CLINICAL TRIAL: NCT00665002
Title: Pilot Trial of a WT-1 Analog Peptide Vaccine in Patients With Myeloid Neoplasms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Innovive Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-15025; INNO-305 WT-1 (Other: Innovive); 105946 (Other: USF IRB)
Record Dates: First submitted 2008-04-18; First posted 2008-04-23 (Estimated); Results first posted 2014-07-24 (Estimated); Last update posted 2015-02-27 (Estimated); Status verified 2015-02

CONDITIONS: Leukemia
Keywords: Myeloid; Monocytic; Hematopoietic; Neoplasms; Acute Myelogenous Leukemia; AML; Myelodysplastic Syndrome; MDS
MeSH Terms: conditions — Leukemia; Neoplasms; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Monatide (IMS 3015); sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- WT-1 Analog Peptide Vaccine (Experimental): Participants received 6 bi-weekly vaccinations over 10 weeks. WT-1 vaccine was given with Montanide. Participants also received an injection of Sargramostim (GM-CSF) two days before each vaccination and again on the day of the WT-1 injection at the same spot.
  Interventions: Biological: WT-1; Drug: Montanide; Drug: Sargramostim (GM-CSF)

INTERVENTIONS:
Biological: WT-1 — Immune responses were to be evaluated at weeks 6 and 12 via delayed-type hypersensitivity, CD4 T cell proliferation, CD4 and CD8 T cell interferon release, as well as by bone marrow cytogenetics including polymerase chain reaction (PCR) to look for molecular evidence of disease. Patients who had an immunologic response and had not had disease progression could continue with up to 6 more vaccinations administered approximately every month. In that case, patients were to be reevaluated with bone marrows/immunologic studies after the 9th and 12th vaccination. In addition, patients would undergo evaluations for residual disease including immunohistochemistry and/or quantitative polymerase chain reaction (RQ-PCR) for WT-1 expression (on selected patients), and multiparameter flow cytometry (AML/ MDS).
  Other Names: Analog Peptide Vaccine
Drug: Montanide — The WT-1 vaccine is given with another substance, called Montanide, which clumps the WT-1 vaccine and thereby improves the immune response.
Drug: Sargramostim (GM-CSF) — GM-CSF was administered at a dose 70 mcg (140ul) as a subcutaneous injection at the site of vaccination on day -2 and day 0.

SUMMARY:
The purpose of this study is to determine whether the WT-1 vaccine causes an immune response and is safe. The WT-1 vaccine is made up of protein pieces that the patient's immune system can recognize as abnormal.

DETAILED DESCRIPTION:
Design:

This will be a pilot trial evaluating the safety and immunogenicity of the WT-1 peptide vaccine in patients with hematologic malignancies. Ten patients with acute myelogenous leukemia (AML) or advanced myelodysplastic syndrome (MDS), will be enrolled. Patients will be vaccinated with a preparation of WT-1-derived native and synthetic peptides plus immunologic adjuvant Montanide ISA 51 VG (Seppic Pharmaceuticals, Fairfield, NJ) and Sargramostim (GM-CSF). One dose level will be tested.

Patients will receive 6 injections of the WT-1 vaccine. Doses will be given every 2 weeks. Each vaccine is given at a different location under the skin in the arm or leg. Patients will be monitored for 30 minutes after vaccination.

WT-1 vaccine is given with another substance, Montanide, which clumps the WT-1 vaccine and improves the immune response. Patients will also receive an injection of Sargramostim (GM-CSF) 2 days before each vaccination and again on the day of the WT-1 injection at the same spot. Sargramostim (GM-CSF) stimulates the body's white blood cells to boost the immune response. Patients may be taught to do the Sargramostim (GM-CSF) injection themselves in which case patients will be given a log sheet to record the injection time and location. If not, they will need to come for an additional 24 study visits.

To monitor their health while receiving the vaccine, patients will need the following tests and procedures as a part of regular cancer care.

* History and physical examination every 2 weeks
* Complete blood count (CBC) and comprehensive panel every 2 weeks
* Bone marrow aspirate at week 14 for patients with acute myelogenous leukemia or myelodysplastic syndrome.

Patients will need these tests and procedures to see whether the vaccine is causing an immune response:

* A skin test will be performed before patients start the study and again in the 8th and 14th weeks in which a small amount of the vaccine will be placed under the skin. Two days later, the site will be checked to see whether a bump or swelling has formed. Another substance which typically does cause a mild reaction (mumps) will also be placed under the skin to measure whether they have a normal immune reaction.
* We will take about 7 tablespoons of blood to measure their immune response. About 1 tablespoon of blood will be taken to measure the levels of WT-1 in their blood. Blood samples will be taken prior to receiving the first vaccination and prior to receiving the vaccination at weeks 6 and 12.

If the vaccine causes the patient to have an immune response, and their cancer does not grow, they may continue to receive the WT-1 vaccinations monthly for 6 more months. If this occurs, the patient will have a computed tomography (CT) scan or bone marrow test and immunology blood tests 2 weeks after the 9th and 12th vaccinations.

ELIGIBILITY:
Inclusion Criteria:

* Cytologic or histologic diagnosis of acute myelogenous leukemia or myelodysplastic syndrome confirmed at Moffitt Cancer Center.
* Patients with acute myelogenous leukemia will have completed induction chemotherapy, achieved first complete remission (CR) 1 or 2, and will have completed any planned postremission therapy (at discretion of treating physician),with no plan for allogenic or autologous transplant.
* Patients with myelodysplastic syndrome who according to the International Prognostic Scoring System (IPSS) are category Int-2 or greater, with disease that relapsed, progressed, or not responded to at least 1 prior course of approved therapy for MDS (i.e. hypomethylating agent or lenalidomide).
* Patients with AML/MDS must have documented WT-1 + disease. For purposes of this study, this may be either the demonstration of WT-1 protein on a pretreatment bone marrow biopsy or detectable disease with RQ-PCR. For patients in whom a bone marrow aspirate is not available or possible (e.g. "dry tap"), a peripheral blood sample may be used for WT-1 screening. In such cases, 10 cc of peripheral blood will be collected in a heparinized tube.
* At least 4 weeks must have elapsed between the patient's last chemotherapy or radiation treatment and the first vaccination.
* Karnofsky performance status ≥ 70%
* Hematologic parameters:

  * Absolute neutrophil count ≥ 1000/mcL (except for MDS, for which the parameter is ≥ 500/mcL)
  * Platelets > 50 K/mcL (except for MDS for which the parameter is > 25 K/mcL and not transfusion dependent)
* Biochemical parameters:

  * Total bilirubin ≤ 2.0 mg/dl
  * Aspartic transaminase (AST) and Alanine transaminase (ALT) ≤ 2.5 x upper limits of normal
  * Creatinine ≤ 2.0 mg/dl

Exclusion Criteria:

* Pregnant or lactating women
* Patients with leptomeningeal disease
* Patients with active infection requiring systemic antibiotics, antiviral, or antifungal treatments
* Patients with serious unstable medical illness
* Patients taking systemic corticosteroids
* Patients with central nervous system (CNS) involvement with cancer/leukemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-06; Primary Completion 2013-07 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Lancet, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- [Derived] Shallis RM, Podoltsev NA. Maintenance therapy for acute myeloid leukemia: sustaining the pursuit for sustained remission. Curr Opin Hematol. 2021 Mar 1;28(2):110-121. doi: 10.1097/MOH.0000000000000637. PMID 33394722

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at Moffitt Cancer Center from 06/30/2008 to 12/13/2012.
Groups:
- Experimental: WT-1 Analog Peptide Vaccine: Participants received 6 bi-weekly vaccinations over 10 weeks. WT-1 vaccine was given with Montanide. Participants also received an injection of Sargramostim (GM-CSF) two days before each vaccination and again on the day of the WT-1 injection at the same spot.
Period: Overall Study
Arm/Group | Experimental: WT-1 Analog Peptide Vaccine
Started | 16
Completed | 4
Not Completed | 12
Not completed — Progression/relapse during treatment | 11
Not completed — Cytogenetic resistance | 1

BASELINE CHARACTERISTICS:
Population: All participants
Arm/Group | Experimental: WT-1 Analog Peptide Vaccine
Number analyzed (Participants) | 16
Age, Continuous [Mean (Full Range); unit: years] | 73 [65 to 82]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: Toxicities were tabulated according to the NCI Common Toxicity (version 3.0) by grade and category. If more than one patient developed ≥ grade 3 non-hematologic toxicity or grade 4 hematologic toxicity, the study accrual was to be suspended immediately for a careful toxicity data evaluation. Depending upon the findings of such safety/toxicity data assessment and consultation with the supporting pharmaceutical company, the principal investigator of this trial would have the option of terminating this trial permanently, amending the study protocol, or resuming the patient accrual.
Time Frame: 12 weeks to 6 months
Population: All participants
Measure: Number; unit: participants
Arm/Group | Experimental: WT-1 Analog Peptide Vaccine
Number analyzed (Participants) | 16
participants | 15

2. Secondary Outcome: Participants Whose Samples Demonstrated Immunological Response After Vaccination
Description: Immune Response: Immune reactivity was measured for all participants. Immune response was measured by T cell proliferative response and DTH against WT-1 peptides. In patients with adequate samples, T cell gamma interferon release as measured by ELISPOT and/or multiparameter intracellular staining by flow cytometry were performed as well.
  ELISPOT Assay: CD4+ immune response, CD4+ and CD8+ response. The samples of participants' blood obtained at baseline and week 12 were tested for CD4 T cell proliferation, CD4 and CD8 T cell interferon release.
  Tetramer Analysis of WT1-specific Immune responses: subtle WT1 T cell expansion, positive by ELISPOT and T cell expansion.
  Delayed-type Hypersensitivity (DTH): measurable DTH response without overlap with ELISPOT or tetramer responders).
  Overall: any form of immune response.
Time Frame: 12 weeks
Population: All participants
Measure: Number; unit: participants
Arm/Group | Experimental: WT-1 Analog Peptide Vaccine
Number analyzed (Participants) | 16
participants
  CD4+ Immune Response | 4
  CD4+ and CD8+ Response | 3
  WT1 T Cell Expansion | 2
  Positive by ELISPOT and T Cell Expansion | 2
  Measurable DTH Response | 2
  Any form of Immune Response | 6

ADVERSE EVENTS:
Time Frame: 4 years, 4 months
Groups:
- Experimental: WT-1 Analog Peptide Vaccine: Participants received 6 bi-weekly vaccinations over 10 weeks.
Arm/Group | Experimental: WT-1 Analog Peptide Vaccine
Serious Adverse Events (participants affected / at risk) | 2/16
Other Adverse Events (participants affected / at risk) | 15/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: WT-1 Analog Peptide Vaccine (N=16)
Gastrointestinal - Other - Appendicitis - unrelated (Gastrointestinal disorders) | 1 (1)
Death Within 100 days - unrelated (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: WT-1 Analog Peptide Vaccine (N=16)
Platelets - low (Blood and lymphatic system disorders) | 10 (16)
Leukocytes (total WBC) - low (Blood and lymphatic system disorders) | 4 (5)
Neutrophils/granulocytes (ANC/AGC) - low (Blood and lymphatic system disorders) | 4 (12)
Hemoglobin - low (Blood and lymphatic system disorders) | 3 (7)
Bone marrow cellularity (Blood and lymphatic system disorders) | 1 (1)
Injection site reaction/extravasation changes (Skin and subcutaneous tissue disorders) | 7 (19)
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 3 (3)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 2 (2)
Rash: erythema multiforme (Skin and subcutaneous tissue disorders) | 2 (3)
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 1 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Flushing (Skin and subcutaneous tissue disorders) | 1 (1)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 8 (10)
Insomnia (General disorders) | 1 (1)
Rigors/chills (General disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (5)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (5)
Anorexia (Gastrointestinal disorders) | 2 (2)
Distension/bloating, abdominal (Gastrointestinal disorders) | 2 (2)
Gastrointestinal - Other (Gastrointestinal disorders) | 2 (2)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 1 (1)
Mucositis/stomatitis (clinical exam) - Anus (Gastrointestinal disorders) | 1 (1)
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Pain - Abdomen NOS (General disorders) | 3 (4)
Pain - Other (General disorders) | 3 (5)
Pain - Bone (General disorders) | 1 (1)
Pain - Head/headache (General disorders) | 1 (1)
Pain - Joint (General disorders) | 1 (3)
Pain - Muscle (General disorders) | 1 (1)
Pain - Neck (General disorders) | 1 (2)
Pain - Sinus (General disorders) | 1 (1)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 2 (2)
Metabolic/Laboratory - Other (Metabolism and nutrition disorders) | 2 (4)
Alkaline phosphatase (Metabolism and nutrition disorders) | 1 (2)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 1 (1)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 1 (1)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Neuropathy: sensory (Nervous system disorders) | 2 (4)
Memory impairment (Nervous system disorders) | 1 (1)
Mood alteration - Anxiety (Psychiatric disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Petechiae/purpura (hemorrhage/bleeding into skin or mucosa) (Blood and lymphatic system disorders) | 2 (2)
Hematoma (Vascular disorders) | 1 (1)
Arthritis (non-septic) (Musculoskeletal and connective tissue disorders) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness, generalized or specific area (not due to neuropathy) Whole body/generalized (Musculoskeletal and connective tissue disorders) | 1 (3)
Dry eye syndrome (Eye disorders) | 1 (1)
Ocular/Visual - Other (Eye disorders) | 1 (1)
Renal/Genitourinary - Other (Renal and urinary disorders) | 1 (1)
Urinary frequency/urgency (Renal and urinary disorders) | 1 (1)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip (Immune system disorders) | 1 (1)
Coagulation - Other (Blood and lymphatic system disorders) | 1 (1)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 (1)
Hot flashes/flushes (Endocrine disorders) | 1 (1)
Edema: limb (Blood and lymphatic system disorders) | 1 (1)
Flu-like syndrome (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes